CLINICAL TRIAL: NCT00397813
Title: Low-Dose TBI Dose Escalation to Decrease Risks of Progression and Graft Rejection After Hematopoietic Cell Transplantation With Nonmyeloablative Conditioning as Treatment for Untreated Myelodysplastic Syndrome or Myeloproliferative Disorders - A Multi-Center Trial
Brief Title: Fludarabine Phosphate and Total Body Irradiation Followed by a Donor Peripheral Stem Cell Transplant in Treating Patients With Myelodysplastic Syndromes or Myeloproliferative Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2056.00; NCI-2010-00237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2056.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Essential Thrombocythemia; Myeloproliferative Neoplasm; Paroxysmal Nocturnal Hemoglobinuria; Polycythemia Vera; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Ring Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Refractory Cytopenia With Multilineage Dysplasia and Ring Sideroblasts
MeSH Terms: conditions — Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Myeloproliferative Disorders; Hemoglobinuria, Paroxysmal; Polycythemia Vera; Primary Myelofibrosis; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm A - Dose Level 1 (Experimental): Arm A - patients with MPD or MDS-RA/RARS Dose Level 1 - 300 cGy TBI
  NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  PBSC TRANSPLANTATION: Patients undergo filgrastim-mobilized PBSC infusion after TBI on day 0.
  IMMUNOSUPPRESSION:
  Matched Related Donor: Patients receive cyclosporine PO BID on days -3 to 56, followed by a taper until day 180. Patients also receive MMF PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.
  Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm A - Dose Level 2 (Experimental): Arm A - patients with MPD or MDS-RA/RARS Dose Level 2 - 400 cGy TBI
  NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  PBSC TRANSPLANTATION: Patients undergo filgrastim-mobilized PBSC infusion after TBI on day 0.
  IMMUNOSUPPRESSION:
  Matched Related Donor: Patients receive cyclosporine PO BID on days -3 to 56, followed by a taper until day 180. Patients also receive MMF PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.
  Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm A - Dose Level 3 (Experimental): Arm A - patients with MPD or MDS-RA/RARS Dose Level 3 - 450 cGy TBI
  NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  PBSC TRANSPLANTATION: Patients undergo filgrastim-mobilized PBSC infusion after TBI on day 0.
  IMMUNOSUPPRESSION:
  Matched Related Donor: Patients receive cyclosporine PO BID on days -3 to 56, followed by a taper until day 180. Patients also receive MMF PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.
  Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm B - Dose Level 1 (Experimental): Arm B - patients with MDS-RAEB or CMML Dose Level 1 - 300 cGy TBI
  NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  PBSC TRANSPLANTATION: Patients undergo filgrastim-mobilized PBSC infusion after TBI on day 0.
  IMMUNOSUPPRESSION:
  Matched Related Donor: Patients receive cyclosporine PO BID on days -3 to 56, followed by a taper until day 180. Patients also receive MMF PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.
  Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm B - Dose Level 2 (Experimental): Arm B - patients with MDS-RAEB or CMML Dose Level 2 - 400 cGy TBI
  NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  PBSC TRANSPLANTATION: Patients undergo filgrastim-mobilized PBSC infusion after TBI on day 0.
  IMMUNOSUPPRESSION:
  Matched Related Donor: Patients receive cyclosporine PO BID on days -3 to 56, followed by a taper until day 180. Patients also receive MMF PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.
  Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm B - Dose Level 3 (Experimental): Arm B - patients with MDS-RAEB or CMML Dose Level 3 - 450 cGy TBI
  NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  PBSC TRANSPLANTATION: Patients undergo filgrastim-mobilized PBSC infusion after TBI on day 0.
  IMMUNOSUPPRESSION:
  Matched Related Donor: Patients receive cyclosporine PO BID on days -3 to 56, followed by a taper until day 180. Patients also receive MMF PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.
  Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo transplantation
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies the side effects and best dose of total-body irradiation when given together with fludarabine phosphate followed by a donor peripheral stem cell transplant in treating patients with myelodysplastic syndromes (MDS) or myeloproliferative disorders (MPD). Giving low doses of chemotherapy, such as fludarabine phosphate, and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. Giving chemotherapy or radiation therapy before or after transplant also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Decrease the incidence of day-200 hematopoietic cell transplantation (HCT) failure to < 20% in patients with MDS-Refractory anemia (RA)-(ringed sideroblasts [RS])/MPD and in patients with chronic myelomonocytic leukemia (CMML)/refractory anemia with excess blasts (RAEB).

SECONDARY OBJECTIVES:

I. The rate of relapse/progression in patients with MPD or MDS-RA and those with CMML or MDS-RAEB.

II. The probability of progression free survival (PFS) in patients with MPD or MDS-RA and those with CMML or MDS-RAEB.

III. The kinetics of donor engraftment.

IV. The incidence of infections.

OUTLINE: This is a dose-escalation study of total body irradiation (TBI).

NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo TBI on day 0.

PERIPHERAL BLOOD STEM CELL (PBSC) TRANSPLANTATION: Patients undergo filgrastim (G-CSF)-mobilized PBSC infusion after TBI on day 0.

IMMUNOSUPPRESSION:

Matched Related Donor: Patients receive cyclosporine orally (PO) twice daily (BID) on days -3 to 56, followed by a taper until day 180. Patients also receive mycophenolate mofetil (MMF) PO BID beginning 4-6 hours after transplantation on day 0 and continue until day 27.

Unrelated Donor: Patients receive cyclosporine PO BID on days -3 to 100, followed by a taper until day 180. Patients also receive MMF PO three times daily beginning 4-6 hours after transplantation on day 0 and continue until day 40, followed by a taper until day 96.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 50 and < 75 years (yrs) with CMML, or previously untreated MDS or MPD
* Patients aged < 50 yrs at high risk for regimen related toxicity using standard high dose regimens; factors considered high risk include pre-existing conditions such as a chronic disease affecting kidneys, liver, lungs, or heart or previous failed HCT
* An human leukocyte antigen (HLA)-identical related or an HLA-matched unrelated donor (Fred Hutchinson Cancer Research Center [FHCRC] matching allowed will be Grade 1.0 to 2.1) is available
* Recovery from the effects of previous chemotherapy, with a minimum of 21 days from initiation of last therapy; hydroxyurea or anagrelide may be used to manage elevated cell counts in patients up to the time they begin therapy under this protocol
* Patients < 12 yrs of age must be discussed on a case by case basis with the primary investigator (PI) of the protocol prior to registration
* A signed informed consent form or minor assent form
* MDS: MDS classifiable by the World Health Organization (WHO) system as RA, RARS, refractory cytopenia with multilineage dysplasia (RCMD), RCMD and ringed sideroblasts (RCMD-RS) or RAEB
* MDS: No previous myelosuppressive therapy; for the purpose of this protocol myelosuppressive chemotherapy will be defined as chemotherapy given with the intent of inducing a complete remission (e.g., standard 7+3, high dose intermittent ARA-C [HIDAC], or Mylotarg)
* MDS: Patients must have < 10% marrow blasts; fewer than 10% marrow blasts must be documented by marrow examination within 3 weeks of initiation of conditioning
* CMML: Patients with CMML1 who have not received myelosuppressive therapy must have < 10% marrow blasts; fewer than 10% marrow blasts must be documented by marrow examination within 3 weeks of initiation of conditioning; OR patients with CMML who have progressed beyond CMML1 and have received myelosuppressive chemotherapy must have < 5% marrow blasts; fewer than 5% marrow blasts must be documented by marrow examination within 3 weeks of initiation of conditioning
* MPD: Patients with polycythemia vera with persistent thrombotic or hemorrhagic complications despite conventional therapy, or who have progressed to postpolycythemic marrow fibrosis
* MPD: Patients with essential thrombocythemia with persistent thrombotic or hemorrhagic complications despite conventional therapy, or who have progressed to myelofibrosis
* MPD: Chronic idiopathic myelofibrosis with peripheral blood cytopenias
* MPD: Patients must have < 10% marrow blasts; fewer than 10% marrow blasts must be documented by marrow examination within 3 weeks of initiation of conditioning
* MPD: No previous myelosuppressive therapy; for the purpose of this protocol myelosuppressive chemotherapy will be defined as chemotherapy given with the intent of inducing a complete remission (e.g., standard 7+3, HIDAC, or Mylotarg)
* Atypical chronic myeloid leukemia (CML): Philadelphia chromosome-negative patients with a diagnosis of atypical CML
* Atypical CML: Patients must have < 10% marrow blasts; fewer than 10% marrow blasts must be documented by marrow examination within 3 weeks of initiation of conditioning
* Atypical CML: No previous myelosuppressive therapy; for the purpose of this protocol myelosuppressive chemotherapy will be defined as chemotherapy given with the intent of inducing a complete remission (e.g., standard 7+3, HIDAC, or Mylotarg)
* Paroxysmal nocturnal hemoglobinuria (PNH): Patients with the non-aplastic form of PNH (cellular bone marrow) who have had a history of life-threatening complications of their disease including thrombotic events, severe hemolysis or Budd Chiari syndrome are eligible; other patients may be considered following approval at PCC and approval by the Principal investigator
* Matched Related Donor: Related to the patient and is genotypically or phenotypically HLA-identical
* Matched Related Donor: Donor age < 75 yrs unless cleared by institutional PI
* Matched Related Donor: Capable of giving written, informed consent
* Matched Related Donor: Donor must consent to PBSC mobilization with G-CSF and apheresis
* Unrelated Donor: FHCRC matching allowed will be grades 1.0 to 2.1: Unrelated donors who are prospectively:

  1. Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing;
  2. Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* Unrelated Donor: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* HLA Matched Related Donor: G-CSF mobilized peripheral blood mononuclear cell (PBMC) only will be permitted as a hematopoietic stem cell (HSC) source on this protocol
* HLA Matched Unrelated Donor: Donor must consent to PBSC mobilization with G-CSF and apheresis; bone marrow unrelated donors are not eligible for this protocol

Exclusion Criteria:

* Organ dysfunction as defined by the following:

  * Symptomatic coronary artery disease or cardiac ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%); if shortening fraction is < 26% a cardiology consult is required with the principal investigator (PI) having final approval of eligibility; ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease
  * Diffusing capacity of the lung for carbon monoxide (DLCO) < 35%, TLC < 35%, forced expiratory volume (FEV)1 < 35% and/or receiving supplementary continuous oxygen; the FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules
  * Liver function abnormalities: Patient with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; the patient will be excluded if he/she is found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, or symptomatic biliary disease
* Bone marrow documenting blast count >= 10% or >= 5% in CMML patients who have progressed beyond CMML1 and received myelosuppressive chemotherapy
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers); this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Presence of >= 5% circulating leukemic blasts (in the peripheral blood) detected by standard pathology
* Active central nervous system (CNS) involvement of disease
* Karnofsky performance score < 70% or Lansky-Play Performance score < 70 for pediatric patients
* Life expectancy severely limited by diseases other than malignancy
* Fungal infections with radiological progression after receipt of amphotericin product or active triazole for > 1 month
* Active bacterial infection
* Patients of fertile age who refuse contraception for a twelve month period post-transplant
* Females who are pregnant or breastfeeding
* Human immunodeficiency virus (HIV) seropositivity
* Severe psychological illness such as major psychosis (e.g. schizophrenia), major bipolar depression, or suicidal situational depression
* Matched Related Donor: Identical twin
* Matched Related Donor: Any contra-indication to the administration of subcutaneous G-CSF at a dose of 16mg/kg/d for five consecutive days
* Matched Related Donor: Serious medical or psychological illness
* Matched Related Donor: Pregnant or lactating females
* Matched Related Donor: Prior malignancy within the preceding five yrs, with the exception of non-melanoma skin cancers
* Matched Related Donor: HIV seropositivity
* Unrelated Donor: A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion; donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results
* Unrelated Donor: Marrow donors
* Unrelated Donor: Donors who are HIV-positive and/or medical conditions that would result in increased risk to the donor G-CSF mobilization and G-PBMC collections
* Unrelated Donor: Serious medical or psychological illness
* Unrelated Donor: Pregnant or lactating females
* Unrelated Donor: Prior malignancy within the preceding five yrs, with the exception of non-melanoma skin cancers
* Unrelated Donor: HIV seropositivity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - LDS Hospital, Salt Lake City, Utah
  - Veterans Administration Center-Seattle, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241
- [Derived] Monaco F, Scott BL, Chauncey TR, Petersen FB, Storer BE, Baron F, Flowers ME, Deeg HJ, Maloney DG, Storb R, Sandmaier BM. Total body irradiation dose escalation decreases risk of progression and graft rejection after hematopoietic cell transplantation for myelodysplastic syndromes or myeloproliferative neoplasms. Haematologica. 2019 Jun;104(6):1221-1229. doi: 10.3324/haematol.2018.199398. Epub 2019 Jan 10. PMID 30630975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
Started | 36 | 0 | 0 | 12 | 5 | 24
Completed | 36 | 0 | 0 | 12 | 5 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3 | Total
Number analyzed (Participants) | 36 | 0 | 0 | 12 | 5 | 24 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 0 | 0 | 5 | 2 | 5 | 30
  >=65 years | 18 | 0 | 0 | 7 | 3 | 19 | 47
Age, Continuous [Median (Full Range); unit: years] | 64.5 [37 to 72] |  |  | 66.5 [58 to 72] | 68 [61 to 69] | 68.5 [53 to 74] | 67 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 |  |  | 7 | 2 | 5 | 24
  Male | 26 |  |  | 5 | 3 | 19 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 35 |  |  | 12 | 4 | 23 | 74
  Unknown or Not Reported | 0 |  |  | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0 | 0 | 0 | 0
  Asian | 0 |  |  | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 | 0 | 0 | 0
  Black or African American | 0 |  |  | 0 | 0 | 0 | 0
  White | 35 |  |  | 12 | 4 | 19 | 70
  More than one race | 0 |  |  | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 |  |  | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 |  |  | 12 | 5 | 24 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With HCT Failure.
Description: HCT failure will be defined as graft rejection (defined as < 5% donor T-cell chimerism) or disease progression within 200 days of transplant.
Time Frame: 200 days
Population: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
Number analyzed (Participants) | 36 | 0 | 0 | 12 | 5 | 24
Participants | 4 | 0 | 0 | 5 | 3 | 2

2. Secondary Outcome: Number of Patients Who Had Infections
Description: Number of patients who experienced bacterial, fungal, or viral infections.
Time Frame: 1 year
Population: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
Number analyzed (Participants) | 36 | 0 | 0 | 12 | 5 | 24
Participants | 24 | 0 | 0 | 12 | 4 | 24

3. Secondary Outcome: Number of Patients Who Engrafted
Description: Continued engraftment will be defined as the detection of donor T-cells (CD3+) as a proportion of the total T-cell of greater than 5%.
Time Frame: 1 year
Population: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
Number analyzed (Participants) | 36 | 0 | 0 | 12 | 5 | 24
Participants | 35 | 0 | 0 | 12 | 4 | 24

4. Secondary Outcome: Number of Patients With Progression-free Survival
Description: Evidence of disease progression will be an indication for therapeutic intervention. Defined as any evidence by morphologic or flow cytometric evaluation of the bone marrow aspirate of an incremental increase in 5% blasts in MDS/CMML; defined as any evidence of blastic transformation in agnogenic myeloid metaplasia/atypical CML; and defined as progressive erythrocytosis, thrombocytosis, or evidence of leukemic transformation in polycythemia vera and essential thrombocythemia.
Time Frame: 1 year
Population: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
Number analyzed (Participants) | 36 | 0 | 0 | 12 | 5 | 24
Participants | 24 | 0 | 0 | 1 | 2 | 11

5. Secondary Outcome: Number of Patients With Relapse/Progression
Description: as for outcome 4
Time Frame: 1 year
Population: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
Number analyzed (Participants) | 36 | 0 | 0 | 12 | 5 | 24
Participants | 6 | 0 | 0 | 6 | 3 | 6

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200; All-Cause Mortality: Conditioning through 1 Year.
Description: No patients were enrolled on arms A2 and A3 because dose escalation was never triggered.
Arm/Group | Arm A - Dose Level 1 | Arm A - Dose Level 2 | Arm A - Dose Level 3 | Arm B - Dose Level 1 | Arm B - Dose Level 2 | Arm B - Dose Level 3
All-Cause Mortality (participants affected / at risk) | 10/36 | 0/0 | 0/0 | 10/12 | 3/5 | 9/24
Serious Adverse Events (participants affected / at risk) | 3/36 | 0/0 | 0/0 | 7/12 | 2/5 | 4/24
Other Adverse Events (participants affected / at risk) | 16/36 | 0/0 | 0/0 | 9/12 | 2/5 | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Dose Level 1 (N=36) | Arm A - Dose Level 2 (N=0) | Arm A - Dose Level 3 (N=0) | Arm B - Dose Level 1 (N=12) | Arm B - Dose Level 2 (N=5) | Arm B - Dose Level 3 (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GVHD (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Psychiatric disorders - Other, specify (altered mental status) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Dose Level 1 (N=36) | Arm A - Dose Level 2 (N=0) | Arm A - Dose Level 3 (N=0) | Arm B - Dose Level 1 (N=12) | Arm B - Dose Level 2 (N=5) | Arm B - Dose Level 3 (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 9 (11) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 6 (6)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 5 (5)
Flu like symptoms (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT00397813/Prot_SAP_000.pdf